CLINICAL TRIAL: NCT01159431
Title: Randomized Double Blind Study of External Trigeminal Nerve Stimulation for Intractable Epilepsy
Brief Title: External Trigeminal Nerve Stimulation for Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Collaborators: Epilepsy Foundation (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Christopher DeGiorgio, PI, Olive View-UCLA Education & Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNS-TDP-01
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Epilepsy; Seizure Disorders
Keywords: partial seizures; poorly controlled epilepsy; intractable epilepsy; treatment resistant epilepsy; Trigeminal Nerve; Trigeminal Nerve Stimulation
MeSH Terms: conditions — Epilepsy; Seizures; Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental)
  Interventions: Device: Trigeminal Nerve Stimulation
- Control (Other)
  Interventions: Device: Trigeminal Nerve Stimulation

INTERVENTIONS:
Device: Trigeminal Nerve Stimulation — External stimulation of the supraorbital branch of the Trigeminal Nerve using a digital TENs unit

SUMMARY:
This study investigates a new therapy for epilepsy called Trigeminal Nerve Stimulation (TNS). TNS involves external electrical stimulation of sensory nerve located above the eyes and over the forehead. The purpose of this study is to determine if TNS is safe and effective using a rigorous randomized active-control clinical trial design in 50 people with epilepsy.

DETAILED DESCRIPTION:
Poorly controlled epilepsy is a disabling condition, affecting over one million Americans. Neurostimulation is a promising alternative for patients who have failed medical therapy, and who are not resective surgical candidates.

Trigeminal Nerve Stimulation (TNS) is a novel form of neurostimulation, and has a strong antiepileptic effect in an animal model of seizures. Preliminary data in humans indicates TNS is well tolerated and may be effective in people with intractable epilepsy.

TNS is an alternative mode of neurostimulation, because the Trigeminal Nerve can be stimulated in minimally-invasive fashion.

This is a randomized double blind study of Trigeminal Nerve Stimulation, which compares high stimulation to an active control. Subjects with poorly controlled partial onset seizures who meet all inclusion and exclusion criteria, enter a 6-week baseline period, and then are randomized in double-blind fashion to high or low intensity stimulation for 18 weeks. 50 subjects are to be enrolled at two sites.

Study outcomes are the following:

1. Percent change in seizure frequency during the treatment period compared with the baseline (pre-treatment) period.
2. Time to the 4th seizure

The primary comparisons will be between and within groups.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 70;
* No serious or progressive medical illness;
* A history of intractable partial seizures;
* At least two complex partial or tonic clonic generalized seizures per month in the last two consecutive months;
* MRI or EEG consistent with localization-related or partial epilepsy;
* Exposure to at least two antiepileptic drugs at adequate doses;
* Concurrent use of at least one antiepileptic drug at adequate doses;
* No change in antiepileptic dose for at least 30 days before study enrollment

Exclusion Criteria:

* History of non-epileptic seizures;
* Inability to maintain accurate seizure calendars (self or caregiver);
* Frequent use of benzodiazepines for clusters defined as greater than four times a month;
* History of facial pain or trigeminal neuralgia;
* Concurrent vagus nerve stimulation;
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M DeGiorgio, MD, Principal Investigator — University of California, Los Angeles; Christi Heck, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - USC Department of Neurology, Los Angeles, California
  - Olive View/UCLA Medical Center, Sylmar, California

REFERENCES:
- [Background] DeGiorgio CM, Murray D, Markovic D, Whitehurst T. Trigeminal nerve stimulation for epilepsy: long-term feasibility and efficacy. Neurology. 2009 Mar 10;72(10):936-8. doi: 10.1212/01.wnl.0000344181.97126.b4. No abstract available. PMID 19273830
- [Result] DeGiorgio CM, Soss J, Cook IA, Markovic D, Gornbein J, Murray D, Oviedo S, Gordon S, Corralle-Leyva G, Kealey CP, Heck CN. Randomized controlled trial of trigeminal nerve stimulation for drug-resistant epilepsy. Neurology. 2013 Feb 26;80(9):786-91. doi: 10.1212/WNL.0b013e318285c11a. Epub 2013 Jan 30. PMID 23365066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited beginning at Olive View/UCLA and Keck-USC between 3/2008 and 10/2010
Pre-assignment Details: 6-week pretreatment baseline
Groups:
- Active: Trigeminal Nerve Stimulation-High Settings
- Control: Trigeminal Nerve Stimulation-Low Settings
Period: Overall Study
Arm/Group | Active | Control
Started | 25 | 25
Completed | 23 | 19
Not Completed | 2 | 6
Not completed — Adverse Event | 1 | 2
Not completed — non-compliance | 1 | 1
Not completed — Lack of Efficacy | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.1 (10.57) | 34.2 (10.81) | 33.44 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 9 | 14 | 23
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: 50% Responder Rate
Description: Change in responder rate, at end of study (18 weeks)
  Absolute percent of subjects with 50% reduction in seizures, 18 weeks compared with 6 weeks Note, the number is not a mean or median, but a fixed percentage.
Time Frame: Treatment period, 18 weeks (end of double blind period) compared with first 6 weeks
Measure: Number; unit: percentage of participants
Groups:
- Treatment: Trigeminal Nerve Stimulation-High Settings
Arm/Group | Treatment | Control
Number analyzed (Participants) | 23 | 19
percentage of participants | 40.5 | 15.6

2. Primary Outcome: Time to the 4th Seizure
Description: Number of Days to the 4th seizure
Time Frame: treatment period (18-weeks)
Measure: Mean (Standard Deviation); unit: days
Groups:
- Control Group-Baseline: Baseline
- Control Group-Double Blind Period: Sham Treatment
Arm/Group | Control Group-Baseline | Control Group-Double Blind Period | Treatment Group-Baseline | Treatment Group-Double Blind Period
Number analyzed (Participants) | 25 | 19 | 25 | 23
days | 23 (19) | 18 (31) | 12.5 (18) | 15 (28)

3. Secondary Outcome: Response Ratio: Mean Percent Change in Seizures
Description: Response Ratio: Mean Percent Change in seizures over the treatment period, where [T-B] / [T+B] x 100%, where T = seizure frequency during the treatment period, and B = seizure frequency during the baseline period.
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: percentage change of RRATIO
Arm/Group | Treatment | Control
Number analyzed (Participants) | 23 | 19
percentage change of RRATIO | -13.9 (6.7) | -9.0 (6.8)

4. Primary Outcome: Change in Seizure Frequency
Description: Percent change in seizure frequency from baseline
Time Frame: 18 weeks
Measure: Median (Standard Deviation); unit: percentage change in seizures per month
Arm/Group | Treatment | Control
Number analyzed (Participants) | 23 | 19
percentage change in seizures per month | -16.1 (15.4) | -10.5 (11.1)

5. Secondary Outcome: Mood
Description: Mean change in score on the Beck Depression Inventory. The Beck Inventory is a patient reported mood scale. The minimum score is 0, and the maximum score is 63. Scores of less than 10 are considered in the normal range. Scores above 10 are consistent with depression. Higher scores indicate higher degrees of depression, with scores of > 25 consistent with severe depression.
Time Frame: 18-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Control
Number analyzed (Participants) | 23 | 19
units on a scale | -8.13 (1.35) | -3.95 (1.22)

ADVERSE EVENTS:
Time Frame: 18-weeks
Description: anxiety
Arm/Group | Active | Control
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 5/25 | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Active (N=25) | Control (N=25)
Seizure cluster (Nervous system disorders) | 0 (0) | 1/24 (1) — Seizure cluster requiring visit to the ER, not device related.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=25) | Control (N=25)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
skin irritation (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
headache (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to sample size and high variability in seizure frequency, median change did not achieve significance. To constrain variability, the RRATIO was used to assess seizure frequency. The RRATIO demonstrated within groups differences, p=0.04 ANOVA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No